CLINICAL TRIAL: NCT05522244
Title: The ExtendeD Computed tomogrAphy angiographY for the successfuL screenInG of Cardioaortic tHrombus in Acute Ischemic Stroke and TIA (DAYLIGHT) Trial
Brief Title: The Extended CTA for the Successful Screening of Cardioaortic Thrombus in Acute Ischemic Stroke and TIA (DAYLIGHT) Trial
Acronym: DAYLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 121385
Record Dates: First submitted 2022-08-17; First posted 2022-08-30 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-04

CONDITIONS: Acute Ischemic Stroke; Transient Ischemic Attack; Intracardiac Thrombus
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard CTA (No Intervention): Standard CTA performed as standard of care for Stroke Workup
- extended CTA (Experimental): The standard CTA will be extended 6 cm below the carina
  Interventions: Diagnostic Test: extended CTA

INTERVENTIONS:
Diagnostic Test: extended CTA — Extending the standard CTA 6 cm below the carina.
  Arms: extended CTA

SUMMARY:
Embolic strokes of undetermined source (ESUS) represent a subset of cryptogenic strokes that are suspected to have an occult embolic source. The risk of stroke recurrence in patients with ESUS varies between 1.9%/year and 19.0%/year depending on the prevalence of vascular risk factors. Part of the elevated recurrence rate is due to the inability to identify high-risk treatable causes such as cardiac thrombi as those found in the left atrial appendage (LAA), left atrium (LA), left ventricle (LV), valves, or aortic arch. The most frequently used diagnostic method in clinical practice to detect cardioaortic thrombi is transesophageal echocardiography (TEE). However, the relatively low availability, higher cost, and invasive nature of TEE limit its large-scale usability. In most stroke centers, patients presenting with an acute ischemic stroke or TIA undergo a tomography (CT) angiography (CTA) of the neck and intracranial vessels. This standard of care CTA (sCTA) classically includes the aortic arch, the higher portion of the ascending/descending aorta, and the rostral portion of the cardiac chambers, but does not involve the LAA, LV, or cardiac valves. A recent study performed among 300 patients with an acute ischemic stroke showed an overall LAA thrombus detection of 6.6% and 15% in patients with AF by extending the CTA 6 cm below the carina. This is an extraordinarily high prevalence of LAA compared to 0.5% to 4.8% of intracardiac thrombi identified on TEE in most previous studies. The major limitation of previous CTA and TEE studies is their observational design, so the differing prevalence of LAA thrombi could be explained by dissimilar population characteristics or selection bias. Based on the methodological limitation of prior studies and the promising role of extended CTAs (eCTA), a randomized controlled trial comparing eCTA + standard of care stroke workup vs. sCTA + standard of care stroke workup is needed.

DETAILED DESCRIPTION:
Between 16% and 25% of patients with ischemic strokes do not have an identifiable cause after a full stroke workup, and their strokes are classified as cryptogenic. Embolic strokes of undetermined source (ESUS) represent a subset of cryptogenic strokes that are suspected to have an occult embolic source. The risk of stroke recurrence in patients with ESUS varies between 1.9%/year and 19.0%/year depending on the prevalence of vascular risk factors. Part of the elevated recurrence rate is due to the inability to identify high-risk treatable causes such as cardioaortic thrombi as those found in the left atrial appendage (LAA), left atrium (LA), left ventricle (LV), valves, or aortic arch.

The most frequently used diagnostic method in clinical practice to detect cardioaortic thrombi is transthoracic echocardiography (TTE). However, the sensitivity of TTE for detecting LV thrombi is as low as 35% without contrast and 64% with proper ultrasound contrast. Furthermore, the sensitivity for LAA thrombi is zero, given that the LAA cannot be visualized on a TTE. Transesophageal echocardiography (TEE) is a better alternative in terms of sensitivity for LV thrombus detection. However, the relatively low availability, higher cost, and invasive nature of TEE limit its large-scale usability.

In most stroke centers, patients presenting with an acute ischemic stroke or TIA undergo a computer tomography (CT) angiography (CTA) of the neck and intracranial vessels. This standard of care CTA (sCTA) classically includes the aortic arch and the higher portion of the ascending/descending aorta, but does not involve the LAA, LV, or cardiac valves. A recent study performed among 300 patients with an acute ischemic stroke showed an overall LAA thrombus detection of 6.6% and 15% in patients with atrial fibrillation (AF) by extending the CTA 6 cm below the carina. This is an extraordinarily high prevalence of LAA compared to 0.5% to 4.8% of intracardiac thrombi identified on TEE in most previous studies. The major limitation of previous CTA and TEE studies is their observational design, so the differing prevalence of LAA thrombi could be explained by dissimilar population characteristics or selection bias. Based on the methodological limitation of prior studies and the promising role of extended CTAs (eCTA), a randomized controlled trial comparing eCTA + standard of care stroke workup vs. sCTA + standard of care stroke workup is needed.

Demonstrating that performing an eCTA can significantly increase the detection of LAA thrombi compared to sCTA has three important implications with the potential to improve clinical practice, patients' outcomes, and clinical guidelines. Furthermore, an eCTA could become part of the standard of care workup of patients presenting to the Emergency Department with a hyperacute ischemic stroke. Proving that eCTA increases the detection of cardio-aortic thrombi in stroke patients in a randomized controlled trial (highest level of evidence) may result in the recommendation of this approach in future guidelines. The increased detection of LAA thrombi may increase the use of oral anticoagulants, which have proven efficacy for the prevention of recurrent strokes in patients with cardiac thrombi, ultimately resulting in fewer stroke recurrences.10 However, proving the latter concept would require a larger randomized clinical trial with stroke recurrence as the primary efficacy endpoint. The LAA is the most frequent source of thromboembolism in patients with AF11 and LAA thrombi are associated with increased detection of AF on cardiac rhythm monitoring, implying that finding an LAA thrombus may help improve the selection of patients who could benefit from prolonged cardiac monitoring after stroke.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with a suspected cerebrovascular event who are evaluated in the Emergency Department or the Urgent Stroke Prevention Clinic at University Hospital, London Health Sciences Centre, London, Ontario, Canada.
* A confirmed diagnosis of stroke or TIA is not mandatory for patient enrollment and randomization. However, patients without a cerebrovascular event will be further excluded from the analysis of efficacy and safety outcomes. Only patients with an adjudicated ischemic stroke or TIA will be included in the latter analyses. The same patient may be included more than once in the study in case of presenting to the hospital with a suspected stroke on different dates. These patients will be excluded only if they had an outcome event (cardioaortic thrombus) previously adjudicated in the study. The reason for including patients more than once is that the cause of the stroke or the stroke mechanism can change with time (e.g. patient with post-stroke MI developing a new LV thrombus, a patient who had a stroke due to AF who is now on anticoagulants and presents with a new contralateral stroke due to severe carotid artery stenosis).

Exclusion Criteria:

* Allergy to iodinated contrast agents
* Pregnancy
* Lack of a peripheral vein access for intravenous contrast administration
* Any contraindication for the clinical use of a CTA for hyperacute stroke care (e.g., end-stage renal disease that contraindicates a CTA), and active or past cancer of the head, neck, or chest)
* Patients with known or newly diagnosed AF will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Outcome: The proportion of participants with a confirmed or "highly suspected" newly diagnosed cardioaortic thrombus | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  The proportion of participants with a confirmed of "highly suspected" newly diagnosed cardioaortic thrombus (LAA, LA, LV, aorta, any aortic branch proximal to the origin of the common carotid or vertebral arteries, valves, or any other cardiac thrombus) after having completed the standard-of-care stroke workup, regardless of a history of AF or newly detected AF. Although the eCTA is extended 6 cm below the carina to target the LAA, cardiac size and position within the mediastinum vary significantly across patients and in most cases, the eCTA will include part of the left ventricle.

SECONDARY OUTCOMES:
Secondary Efficacy Outcome 1: The proportion of participants diagnosed with a cardio-aortic embolic source that has an available guideline-supported treatment including thrombi, vegetations, and tumors. | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  The proportion of participants diagnosed with a cardio-aortic embolic source that has an available guideline-supported treatment including thrombi, vegetations, and tumors. This outcome does not include other cardio-aortic embolic sources with a guideline-supported treatment that are primarily detected by TTE (part of the standard of care workup in stroke patients) such as high-risk PFO in young patients, acute anterior myocardial infarction with reduced ejection and no LV thrombus fraction (American Heart Association -AHA Guidelines)14, severe LV dysfunction with ejection fraction ≤35%, without evidence of LA or LV thrombus in (Canadian Secondary Prevention Best Practice Recommendations).
Secondary efficacy outcome 2: The proportion of participants diagnosed with a cardio-aortic embolic source known to increase the risk of stroke. | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  The proportion of participants diagnosed with a cardio-aortic embolic source known to increase the risk of stroke. This category includes the following cardio-aortic embolic sources:
  * Any of the components of the primary efficacy outcome.
  * Non-thrombotic slow LAA flow (SLAAF)
  * Moderately to severely enlarged LA (≥42 ml/m2).
  * Reduced LV ejection fraction <35%.
  * High-risk PFO (either a mobile/aneurysmal atrial septum or ≥20-bubble right-to-left shunt) in individuals ≤60 years of age or in older individuals with evidence of venous thromboembolism (pulmonary embolism or deep vein thrombosis).
  * Apical aneurysm/hypokinesis/akinesis, anterior wall hypokinesis/akinesis, or global hypokinesis/akinesis.
  * High-risk aortic plaque defined as >4 mm thickness
  * Aortic dissection involving the aortic arch, ascending, or descending26 aorta.
Secondary efficacy outcome 3: The proportion of participants diagnosed with a cardio-aortic embolic source resulting in the initiation of a new secondary prevention treatment other than antiplatelet therapy. | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  The proportion of participants diagnosed with a cardio-aortic embolic source resulting in the initiation of a new secondary prevention treatment other than antiplatelet therapy, including anticoagulation, antibiotic therapy for infective endocarditis, completed or planned surgery for vegetations in infective endocarditis or aortic dissection, statin therapy in the presence of severe aortic plaque, etc. Initiation of a new therapy will be defined as a treatment started after the stroke, which the participant was not receiving before the stroke occurrence.

OTHER OUTCOMES:
Tertiary efficacy outcome 1: Detection of a pulmonary nodule or mass. | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  Detection of a pulmonary nodule or mass measuring ≥ 6mm, multiple nodules of any size, or a pulmonary mass, as per the Fleischner Society 2017 Guidelines for Management of Incidentally Detected Pulmonary Nodules in Adults.
Tertiary efficacy outcome 2: The detection of pulmonary embolism. | After having complete the standard of care stroke workup for the qualifying stroke or TIA.
  The detection of pulmonary embolism.
Tertiary efficacy outcome 3: Association between Slow LAA Flow and Cognitive Impairment in Stroke Patients. | Through study completion, an average of 1 year
  Association between Slow LAA Flow and Cognitive Impairment in Stroke Patients. Slow flow in the left atrial appendage (LAA) serves as a marker of left atrial cardiopathy, which has been suggested to have implications in the pathogenesis of dementia. Our study aims to examine the potential link between slow LAA flow and cognitive impairment in individuals with a history of stroke.
Primary Safety Outcome 1: door to sCTA time vs door to eCTA | Through study completion, an average of 1 year
  Door-to-CTA completion will be measured to ensure that the eCTA will not result in substantial delays in patient care. Although we anticipate that the eCTA will only be 3 seconds longer than the sCTA, we will aim to document any possible differences.
Secondary Safety Outcome 1: Door-to-needle | Through study completion, an average of 1 year
  Door-to-needle time in patients receiving intravenous thrombolysis is defined as the time elapsed between patient registration at the Emergency Department and the initiation of tPA or TNK bolus.
Secondary Safety Outcome 2: Door-to-groin puncture | Through study completion, an average of 1 year
  Door-to-groin puncture time in patients undergoing mechanical thrombectomy.
Secondary Safety Outcome 3: CTA-related radiation exposure | Through study completion, an average of 1 year
  Radiation exposure will be retrieved from the CTA summary report, which is reported as Dose Length Product (DLP) in milligray-centimeter (mGy-cm). The DLP is reported separately for the body and head. Each measure will be multiplied by their respective dose conversion coefficients (k factors), which account for the radiosensitivity of organs in the scanned region, to estimate the effective dose reported in millisievert (mSv).
Secondary Safety Outcome 4: Contrast-induced nephropathy | Through study completion, an average of 1 year
  Contrast-induced nephropathy, defined as an increase in serum creatinine ≥44 µmol/L (0.5 mg/dL) or a 25% increase from baseline within 48 hours after contrast exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Sposato, MD, Principal Investigator — London Health Sciences Center, Western University; Rodrigo Bagur, MD, Principal Investigator — London Health Sciences Center, Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Sposato LA, Ayan D, Ahmed M, Fridman S, Mandzia JL, Elrayes M, Lodol F, Khaw AV, Mai LM, Bogiatzi C, Casserly C, Fraser JA, Chan R, Florendo Cumbermack A, Markovic N, Yu Y, Debicki D, Fleming L, Beauchamp B, Lambourn L, Mayich M, Milroy L, Sharma M, Pandey S, Bagur R. Extended CT angiography versus standard CT angiography for the detection of cardioaortic thrombus in patients with ischaemic stroke and transient ischaemic attack (DAYLIGHT): a prospective, randomised, open-label, blinded end-point trial. Lancet Neurol. 2025 Jun;24(6):489-499. doi: 10.1016/S1474-4422(25)00111-5. PMID 40409313